CLINICAL TRIAL: NCT06770816
Title: Effect of Left Erector Spinae Plane Block on Left Ventricular Functions
Acronym: ESP-LV ECHO
Status: Not yet recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, ass. prof.dr, Aydin Adnan Menderes University
Other Study IDs: 221
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Erector Spina Plan Block; Echocardiography
Keywords: erector spina plan block; left ventricle; echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- erector spina plan block: ESP block will be applied from the midline 3 cm lateral to the T5 level under ultrasound guidance. After the area is cleaned with povidone iodine before the block, the T5 transverse process will be determined using a linear ultrasound probe. Local anesthetic will be applied between the transverse process and the erector spinae muscle with the help of an insulated needle designed for peripheral block procedures. The location of the needle will be verified with the hydrodissection method with physiological serum without local anesthesia. After the location of the needle is verified, 0.25% bupivacaine 20 ml mixture will be applied.
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — HR, MAP, SBP and DBP will be recorded at baseline and 15 minutes after ESP block. Cardiac output (CO) will be calculated using echocardiographic data on stroke volume (SV) (measured from the LV outflow tract) and multiplied by HR. Changes in LV systolic function will be assessed with three parameters: fractional shortening (FS), ejection fraction (EF) using the Simpson method and S' wave of tissue Doppler imaging (TDI) of the mitral annulus (average of values at the medial and lateral annulus). LV diastolic function will be assessed with three parameters and interpreted according to the European Association of Cardiovascular Imaging guidelines. Pulsed wave (PW) Doppler of trans-mitral flow will be used to obtain the ratio between early (e) and late (atrial, a) waves. A PW Doppler between the LV outflow tract and the mitral valve will be performed to estimate the iso-volumetric relaxation time IVRT. TDI will be used to investigate myocardial relaxation at the mitral annular level (ear

SUMMARY:
Many studies have shown a decrease in inotropic status (intrinsic function) after blockade of cardiac sympathetic innervation with thoracic epidural anesthesia (TEA) (4,5). There is no study in the literature investigating the cardiac effects of left thoracic ESP block. We think that left thoracic ESP block, like TEA, may also have cardiac effects. Therefore, we aimed to investigate the effect of left thoracic ESP block on left ventricular functions with transthoracic echocardiography (TTE).

DETAILED DESCRIPTION:
After extubation, respiratory therapy and pain management are important issues in postoperative care. Adequate postoperative pain control is necessary for a good respiratory effort. For years, the use of intravenous opioids has become the standard in pain management. Opioids administered to adequately control pain may cause sedation and respiratory depression. Due to the large number of opioid-related side effects, alternative pain relief methods are being sought.

Erector spinae area (ESP) block has recently been described in the treatment of pain after thoracic surgery (1,2,3).

The focus of this section is left thoracic ESP block, in which the cardiac sympathetic nerves (T1-T5) are involved in neural blockade. Many studies have shown a decrease in inotropic status (intrinsic function) after blockade of cardiac sympathetic innervation with thoracic epidural anesthesia (TEA) (4,5). There is no study in the literature investigating the cardiac effects of left thoracic ESP block. We think that left thoracic ESP block, like TEA, may have cardiac effects. Therefore, we aimed to investigate the effect of left thoracic ESP block on left ventricular functions with transthoracic echocardiography (TTE).

The study was designed as an observational study. After obtaining written informed consent from the patients, it was planned to apply the routine ultrasonography-guided ESP block to the patients. This application is performed in thoracic surgeries performed with general anesthesia as standard in our hospital.

Demographic data to be obtained, in addition to the outcomes of the above-mentioned study, will include recording height (cm), weight (kg), age (years), gender, (ASA) physical condition, and specific procedure type. Patients will be asked about tobacco and alcohol use, drug use. They will also be asked about their medical history, including lung disease, kidney disease, diabetes mellitus, neurological disease, chronic pain conditions, previous surgery or stent placement, and medications. Current preoperative laboratory tests and medication list will be recorded. Parameters measured by TTE before and 15 minutes after the block will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective left-sided thoracic surgery ASA I-III 18-75 years of age

Exclusion Criteria:

1. Refusal at enrollment
2. Request for withdrawal from the study
3. Inability to give informed consent
4. Emergency surgery
5. Bleeding diathesis
6. Presence of contraindications to the LA agents used in this study
7. Use of chronic opioids
8. Psychiatric disorders
9. Presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo elective left-sided thoracic surgery, ASA I-III and between the ages of 18-75
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic assessment of left ventricular function | Left ventricular function will be assessed by echocardiography 15 minutes before and 15 minutes after left high thoracic esp block.
  Standard measurements of left ventricular systolic function include left ventricular volumes (indexed to body surface area, BSA), left ventricular ejection fraction (LVEF) according to the modified Simpson rule, time and velocity integral in the left ventricular outflow tract (TVI-LVOT), and stroke volume (SV) (= π x LVOT radius2 x TVI-LVOT). Stroke volume index (SVI) will be calculated as SV/BSA. Mitral and aortic Doppler flow profiles, left ventricular isovolumetric relaxation time, and maximum flow velocity measurements will be recorded. LV early (E-max) and late (A-max) diastolic filling will be assessed.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Missant C, Claus P, Rex S, Wouters PF. Differential effects of lumbar and thoracic epidural anaesthesia on the haemodynamic response to acute right ventricular pressure overload. Br J Anaesth. 2010 Feb;104(2):143-9. doi: 10.1093/bja/aep354. Epub 2009 Dec 22. PMID 20031952